CLINICAL TRIAL: NCT01784783
Title: HIV Testing and Educating Male Partners to Improve Maternal and Infant Outcomes: Home-based Partner Education and Testing (HOPE) Study
Brief Title: Home-based Partner Education and Testing (HOPE) Study
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carey Farquhar, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 44357-A; R01HD075108-01 (NIH)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: HIV
Keywords: HIV transmission; PMTCT; Discordancy; Home-based testing; Couple counseling; Couple testing; Facility delivery; Exclusive breastfeeding; Family planning; Postpartum contraceptives; Linkage to care; ART initiation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOPE Intervention (Experimental): Pregnant women and their male partners will receive home-based couple HIV testing and counseling and partner education 1-2 weeks after enrollment. The intervention will include educational messages concerning socio-behavioral, condom-based, and treatment-oriented approaches to prevention of horizontal and vertical HIV transmission, based on the status of each of the partners. The couple will also be educated about the importance of facility delivery, exclusive breastfeeding, family planning, and post-partum contraception.
  During the HOPE Intervention, the purpose and design of the study will be explained to male partners. Men will be asked to provide written informed consent for study participation. Provided they consent, men will complete a questionnaire asking for sociodemographic characteristics, medical and sexual history, behavioral data and information on prior HIV testing and counseling.
  Interventions: Behavioral: HOPE Intervention
- INVITE Intervention (Experimental): Pregnant women will be tested and encouraged to bring their male partners to the antenatal clinic for testing. Women will receive a clinic invitation to give to their male partners to attend the next visit for couple HIV counseling and testing. The couples will also be offered the relevant components of the intervention at the final study visit, 6 months postpartum.
  Interventions: Behavioral: INVITE Intervention

INTERVENTIONS:
Behavioral: HOPE Intervention — If the male partner chooses not to complete the study questionnaire, he may decline and participate only in the HOPE intervention component of the study. (This does not preclude the possibility of the female partner continuing to participate in the study.) Investigators anticipate that this will occur and also expect that some women and male partners randomized to the intervention arm will refuse the HOPE intervention when offered. Study staff will attempt to collect data on reasons for refusal to participate and will continue to follow these couples through 6 months postpartum to collect maternal and infant outcome data, provided the female partner does not withdraw from the study.
  Key educational messages will be presented using an electronic tablet highlighting key messages and will include with relevant images as visual aids. This will help to facilitate comprehension and ensure that all relevant materials are covered during each intervention session.
  Arms: HOPE Intervention
Behavioral: INVITE Intervention — Women will receive a clinic invitation to give to their male partners to attend the next antenatal visit for couple HIV counseling and testing.
  Arms: INVITE Intervention

SUMMARY:
The purpose of this study is to investigate the impacts of home-based couple HIV-testing and counseling and male partner education on partner HIV testing and other critical maternal and infant health outcomes during pregnancy and the postpartum period. Additionally, the study seeks to assess the cost-effectiveness of this approach.

Involvement of men during the antenatal and postpartum period, including HIV testing of male partners, can have substantial benefits for women and infants. In observational studies, male participation in antenatal care has been associated with increased uptake of prevention of mother-to-child transmission (PMTCT) interventions, and more recently, a study in Kenya found a significant HIV-free survival benefit for children of HIV-infected women whose male partners attended antenatal care where couple HIV testing was offered. In this study only 31% of ~450 men invited for counseling and testing came to clinic, highlighting the challenges faced across sub-Saharan Africa when trying to access male partners of pregnant women.

In areas of high HIV-1 prevalence, high levels of male involvement may be readily achievable because home-based counseling and testing is highly acceptable and the benefits of male participation and HIV testing extend to HIV-uninfected pregnant and postpartum women and infants. Reaching out to men during pregnancy may reduce incident HIV infection and vertical transmission among these women, but efforts to engage men in antenatal care in Western Kenya have thus far achieved limited success. This intervention may achieve gains beyond prevention of maternal and infant HIV-1 acquisition through identification of HIV-infected men who would otherwise not learn their status or delay treatment, and by improving child health through targeted education of male partners. When administered in a home-based setting simple, established interventions such as the promotion of exclusive breastfeeding have been shown to be associated with significant reductions in child mortality. Home-based approaches also lend themselves to integration with targeted interventions such as promotion of HIV testing among male partners of at-risk pregnant women. Furthermore, a successful HIV testing program for male partners of pregnant women has potential to reach a large number of men who may be unaware of their HIV status or who are HIV-infected but not in care, providing linkages to treatment clinics and promoting prevention interventions, such as safe sex and voluntary male circumcision for those who are uninfected.

In this randomized clinical trial up to 600 couples (300 in each treatment arm) will be randomized to standard antenatal care or home-based partner education and HIV testing (HOPE) as part of routine pregnancy services. Women will be enrolled at the antenatal clinic in Kisumu District Hospital, Kisumu, Kenya. Couples in the control group will receive the HOPE Intervention, featuring home-based couple counseling and HIV testing as well as key educational messages concerning HIV prevention behaviors, facility delivery, exclusive breastfeeding, and post-partum family planning. Women in the control arm will be invited to bring their male partners to the antenatal clinic for voluntary clinic testing and counseling. Women will be followed up at clinic visits 6-weeks and 14-weeks postpartum and again with their male partner 6-months post-partum. These follow-up visits will include questionnaires to measure uptake of HIV testing, facility delivery, exclusive breastfeeding and postpartum contraceptive use as well as linkage to HIV care. Cost-effectiveness of the intervention will also be evaluated in order to inform future scale-up.

First, the investigators hypothesize that successful implementation of HOPE will result in higher uptake of male partner HIV testing, couple testing and disclosure of HIV status. The investigators also hypothesize that there will be benefits to HIV-infected and HIV-uninfected women and their children who will have improved uptake of interventions to improve maternal and child health. Specifically, the investigators anticipate higher levels of facility delivery, optimal breastfeeding practices, and post-partum contraceptive use, as well as increased uptake of antiretroviral treatment for HIV+ women in the intervention arm, relative to the control arm. Second, the investigators hypothesize that greater than 85% of HIV-1-infected men identified through home-based partner education and testing (HOPE) will access care and treatment services, and, overall, more women in the HOPE arm will know their partners' status at each time point and more partners will be in care and treatment. Third, the investigators predict that uptake of counseling and testing and HIV prevalence among male partners and family members will be high enough to make this approach cost-effective from both payer and societal perspectives.

DETAILED DESCRIPTION:
1. Study design:

   The proposed study is a randomized clinical trial to determine the effect of offering home-based partner education and testing (HOPE) to pregnant women. Up to 600 women will be enrolled and randomly assigned to the HOPE intervention (home-based partner education and testing - HOPE) and INVITE arms (clinic invitation to male partner to attend couple HIV counseling and testing). Women will be recruited into the study when they present for routine antenatal care.
2. Study Area Description:

   This proposed trial will be carried out in and around Kisumu, located in Western Kenya, in collaboration with Kisumu District (now County) Hospital. This site has been selected because it has a high volume of new antenatal visits (~200/month), and high HIV prevalence among women presenting for antenatal care (~9.5-12%), which correlates with high HIV-1 incidence in this population. This will enable us to achieve the necessary number of outcome events in the desired timeframe. Kisumu District Hospital provides HIV testing to women and couples and offers PMTCT interventions to pregnant and postpartum HIV-1-infected women according to the Kenya Ministry of Health guidelines, which include ART when indicated. The facility adheres to the Kenyan national infant feeding policy and provides infant feeding counseling for pregnant and lactating women and their partners, emphasizing the benefits of breastfeeding and advocating for exclusive breastfeeding during infants first 6 months of life.
3. Sample Method:

   Women will be recruited at the antenatal clinic at Kisumu District Hospital. All consenting women who report for care at the clinic will be screened, and all who are eligible will be invited to participate (continuous enrollment).
4. Recruitment:

   Women will present to the antenatal clinic at Kisumu District Hospital, at which point they will be introduced to the study by study nurses and verbally asked for permission to be screened for eligibility. (A waiver of written consent is requested for screening.) Women who agree will be screened for eligibility, and eligible women will be invited to complete the consent process and provide written consent as a prerequisite for participation in the study. Scripts regarding information about the study and invitation to the study, which will be used by study nurses, are included in the screening forms, found in the appendix.

   Male partners will be approached at a home locator visit (a telephone call will be made if the man is not present), at which point the study's health advisors will introduce the study to the men. Men will be asked for permission to be screened for eligibility (waiver of written consent). Men who agree will be screened for eligibility and eligible men will be invited to the study and go through the consent process (written consent). Scripts regarding information about the study and invitation to the study, which will be used by study health advisors, as well as home visit and telephone contact protocols are included in the enrollment forms, found in the appendix. It is expected that some men will decline participation, and, although male partner participation is an important component of the study, male enrollment is not a prerequisite for the enrollment and continued participation of their female partners.
5. Enrollment:

   Eligible women recruited at the Kisumu District Hospital Antenatal Clinic will be invited to the study and go through the consent process (written consent). Women will be invited to enroll the same day as they are screened. However, those who desire more time to consider their potential participation will be offered the option of returning the next day to enroll in the study. Once enrolled, women will be interviewed with a standardized questionnaire and tested for HIV using a HIV-1 rapid test. All women will have a home visit to verify and record the location of their home using GPS technology within 1 week of enrollment, as this will help to ensure follow-up in later stages of the study.
6. Randomization:

   This study is a randomized clinical trial. At the end of the enrollment visit, women will be randomized to the HOPE treatment or the INVITE arm based on computer-generated block randomization.
7. Consent Procedure:

   During screening, women will be asked for verbal consent during the screening process, and they will be presented with a consent form and asked for written consent at their enrollment visit. Men will be offered the consent form during the home visit or HOPE intervention. Participants can opt out of the study at any time.
8. Data Collection Procedure:

   A. Basic details:

   Women in both study arms will have a clinic enrollment visit, two clinic visits postpartum at 6 and 14 weeks which correspond with childhood immunization visits, and a home visit at 6 months postpartum. Participants will be reimbursed at 300 Kenyan shillings per clinic visit and 200 Kenyan shillings per home visits. Irrespective of treatment status (i.e. standard ANC or HOPE arm), women will receive a home visit for tracing and retention purposes within 1 week of enrollment and one home visit at the end of follow-up when women are 6 months postpartum. Women in the intervention arm will have an additional home visit for home-based counseling and testing which will occur within 1-2 weeks of enrollment. Each of these visits is described below in more detail and outlined in the study design flowchart.

   B. Enrollment visit:

   In addition to provision of informed consent and randomization, women in both arms will be interviewed and examined. Peripheral blood specimens will be collected for HIV-1 rapid testing, and questions will be asked about demographic and socio-behavioral characteristics, medical, sexual, and reproductive history, and any recent or current symptoms. All women will then be asked to allow a counselor on the study team to accompany them home to confirm locator information for future tracing and retention efforts.

   C. Home visit:

   All women in the proposed study will have a home visit to confirm the physical location of the their home because written addresses are often unreliable. For our mother-to-child HIV transmission studies and HIV-discordant couple studies in Kenya, conducting a home visit on the day of enrollment or shortly thereafter has been highly acceptable and a critical component of an effective tracing and retention plan. Among HIV-discordant couples in Dr. Farquhar's recent prospective cohort study, uptake of the home visit was 97% and for pregnant HIV-infected women in Nairobi, the proportion agreeing to home visit also exceeded 95%. For this study, a written description of the physical location will be recorded by the counselor visiting the woman, and this will be incorporated into the woman's study file in addition to GPS coordinates, recorded using handheld devices that have been used successfully in Nairobi and other regions in Kenya by this research group. During the home visit, male partners of women randomized to the HOPE intervention will be asked to discuss their availability for the HOPE intervention when community health workers will next return. Alternatively, if the male partner is not at home, he will be contacted via phone or home visit to schedule a return visit.

   D. Intervention and control arm procedures:

   (See Interventions section)

   E. Postpartum follow-up visits:

   Three postpartum follow-up visits will occur in the clinic at 6 and 14 weeks postpartum when women return with their infants to receive routine immunizations and at 6 months postpartum at home. At these visits, women will complete a brief questionnaire, and blood will be drawn for rapid HIV testing at the 6-month visit.
9. Retention procedures:

   Retention and tracing will be high priorities in this study. By design, there are only two follow-up visits prior to the 6-month final visit because more frequent follow-up with rapid HIV testing of women could alter women's behavior and reduce the observed effect of the home-based partner education and testing (HOPE) intervention. To minimize loss to follow-up, study staff will perform home visits for participants in both treatment arms and ask for at least 3 phone numbers of people who could be contacted if the participant is not responding to calls. In past studies these two approaches have been extremely effective for tracing individuals and couples. Additionally, active tracing will begin two weeks after the missed visit, for any women not presenting for their visits at 6-weeks or 14-weeks postpartum.
10. Diagnosis and treatment of incident HIV-1 infection among women:

    For women who are initially HIV-seronegative, results of the 6-month rapid HIV tests will be provided as soon as they are available, and women with incident infection will be referred for initiation of antiretroviral treatment (ART). Study clinics and referral clinics will be educated about the importance of rapid initiation of ART when a woman is newly infected to promote immediate treatment. As a result of this education and given existing standard of care practices, sites will be prepared to provide ART at the study clinic and ensure that ART is initiated. When available, existing on-site PMTCT programs will be utilized to leverage PEPFAR and government resources and procure drugs for HIV-infected women at these sites. However, since national supplies may be inconsistent, the study team is prepared to supplement these stocks.
11. Diagnosis, treatment, and follow-up of HIV-1 infection in male partners:

    In the regions surrounding Kisumu HIV-1 seroprevalence among women is estimated to be between 10-15%. Assuming a fairly substantial level of male participation (>75%), investigators anticipate diagnosing upwards of 25 men with HIV infection during the partner testing intervention. These men will be referred to the nearest Comprehensive Care Clinic (CCC) for CD4 testing, HIV care, and ART if indicated. For Aim 3, uptake of HIV care and treatment services among men testing HIV-seropositive during home-based testing will be measured using self-reports from the home visit at 6 months postpartum. A questionnaire will be used to assess the following outcomes: 1) presentation to the CCC for counseling, 2) initiation of trimethoprim-sulfamethoxazole, 3) acceptance of CD4 testing, and 4) ART initiation among those men who are eligible. While the study clinic does not anticipate needing to provide ART for these men, efforts will be made to ensure rapid uptake of ART by men identified as being at high-risk for transmitting HIV-1 to their female partners. The clinic will provide ART if necessary to bridge periods when medications are not available.
12. Provision of services for intimate partner violence:

    While there does not appear to be an increased risk of intimate partner violence (IPV) associated with HIV testing, IPV is common among women in Africa and was considered in the design and implementation of this study. Investigators will monitor IPV by measuring it at enrollment and at each follow-up visit. Women reporting IPV will be encouraged to utilize counseling and education services, and counselors will be made available.
13. Laboratory procedures:

Infant filter paper assays will be performed on-site in the Kisumu KEMRI/CDC Laboratory which is located in close proximity to the study clinic. Study motorcycles will be used to transport specimens. HIV-1 rapid testing will be performed as part of routine care provided in the study clinics. Current protocols in the Kenyan national Voluntary Counseling and Testing (VCT) guidelines specify use of two commercial kits that are locally available, the Determine® HIV-1/2 Rapid Test (Abbott Laboratories) and the Uni-GoldTM Recombigen HIV Test (Trinity Biotech). Infant filter paper specimens will be assayed for HIV-1 DNA using PCR at the Kisumu KEMRI/CDC Laboratory following established protocols and Kenya national guidelines for infant testing.

ELIGIBILITY:
Inclusion Criteria:

Females:

* > 8 weeks gestation
* ≥ 14 years old (all pregnant females 14-17 years old are emancipated minors per Kenyan law)
* Current stable partnership (married or cohabiting)
* Planning on living in vicinity (approx. 40 km or less from clinic) for 9 months postpartum
* Willing to be randomized to intervention or standard of care
* Willing to participate in couple HIV testing and counseling
* No recent history of intimate partner violence (within last month with their current partner)
* Male partner not present during screening visit

Males:

* ≥ 18 years old
* Willing to participate in couple HIV testing and counseling

Exclusion Criteria:

Females:

* ≤ 8 weeks gestation
* < 14 years old (all pregnant females 14-17 years old are emancipated minors per Kenyan law)
* Not in a current stable partnership (not married or not cohabiting)
* Not planning on living in vicinity (approx. 40 km or less from clinic) for 9 months postpartum
* Recent history of intimate partner violence (within last month with their current partner)
* Unwilling to be randomized to intervention or standard of care
* Unwilling to participate in couple HIV testing and counseling
* Male partner present during screening visit

Males:

* < 18 years old
* Unwilling to participate in couple HIV testing and counseling

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Male self-report of uptake of HIV testing | 6 months postpartum
  For both arms, male partners will be asked to report whether they received HIV testing during the course of the study.

SECONDARY OUTCOMES:
Female self-report of delivery location | 6 weeks postpartum
  Female participants will be asked to report where they delivered their baby (e.g. health facility, home, family member's home).
Female self-report of delivery assistance | 6 weeks postpartum
  Female participants will be asked to report who assisted them during delivery (e.g. doctor, nurse, traditional healer, midwife, mother-in-law, etc.)
Female self-report of exclusive breastfeeding | 6 weeks, 14 weeks, and 6 months postpartum
  Female participants will be asked whether they are currently breastfeeding exclusively.
Female self-report of introduction of foods other than breastmilk | Delivery date to 6 weeks, 14 weeks, and 6 months postpartum
  Female participants will be asked when milk substitutes (i.e. formula, cow milk) or other foods were introduced to their child.
Self report of number of sexual partners (female and male) | Enrollment and 6 months postpartum
  Men and women (at enrollment and/or 6 months postpartum) will be asked to report the number of sexual partners they have had during the previous 6 months.
Male self-report of male condom use | Enrollment and 6 months postpartum
  Male participants will be asked to assess their level of condom use during sexual intercourse since during the previous 6 months. Options include 1) always, 2) most occasions, 3) rarely, and 4) never.
Female self-report of date of first receptive intercourse after delivery | 6 weeks, 14 weeks, and 6 months postpartum
  At each follow-up visit, women will be asked whether they have resumed receptive sexual intercourse and, if so, the general time frame that they resumed sex. Upon reporting that they have resumed sexual activity they will no longer be asked this question at remaining interviews.
Female report of male condom use | Enrollment to 6 weeks, 14 weeks, and 6 months postpartum
  Female participants will be asked to assess their partner's level of condom use during sexual intercourse in the previous 6 months (at enrollment and 6 months postpartum) and/or since the last study interview. Options include 1) always, 2) most occasions, 3) rarely, and 4) never.
Self-report of condom use during last sexual intercourse (male and female) | Enrollment, 6 weeks postpartum, 14 weeks postpartum, 6 months
  At each study interview, participants will be asked if they used condom the last time they participated in sexual intercourse.
Female self-report of contraceptive use | 6 weeks, 14 weeks, 6 months postpartum
  After reporting having resumed sexual activity, women will be asked whether they are using contraception. If so, they will be asked what type of contraceptive they have used and how often (for oral medication) or when (for an injectable) they last utilized the contraceptive.
Awareness of partner HIV-status | 6 months postpartum
  Male and female subjects in both the intervention and control arm will be asked to report if they know their partner's status and whether their partner is HIV-negative or HIV-positive.
Awareness of partner HIV status (intervention arm) | Enrollment to 6 months postpartum
  Subjects randomized to the intervention arm will be asked to identify their partner's HIV status during enrollment and at 6 months postpartum. The difference between awareness of partner HIV status before and after the intervention will be evaluated.
Male self-report of linkage to HIV care | 6 months postpartum
  Men who tested HIV-seropositive during the study will be asked to report whether they presented to the Comprehensive Care Clinic.
Male self-report of linkage to HIV care for CD4 testing | 6 months postpartum
  Men who tested HIV-seropositive during the course of the study will be asked to report whether they received CD4 testing at the Comprehensive Care Clinic.
Male self-report of ART initiation | 6 months postpartum
  HIV-positive male partners will report whether they initiated ART and if not, whether they are eligible.
Male self-report of adherence to antiretroviral treatment | 6 months postpartum
  Men who report initiation of ART will be asked report on their degree of adherence to ART on a visual analogue scale.
Female self-report of initiation of prophylaxis | 6 weeks postpartum
  HIV+ Women will report whether they initiated prophylaxis.
Female self-report of Nevirapine treatment for infants | 6 weeks, 14 weeks, 6 months postpartum
  HIV+ women who reported initiating prophylaxis will be asked whether their infants initiated Nevirapine treatment regimens.
Female report of infant adherence to Nevirapine | 6 weeks, 14 weeks, and 6 months postpartum
  Women who reported infant initiation of Nevirapine will be asked report the degree of the infants adherence to the regimen on a visual analogue scale.
Female self-report of initiation of antiretroviral treatment | Enrollment to 6 weeks, 14 weeks, and 6 months postpartum
  ART-eligible, HIV-positive pregnant subjects will be asked to report whether they initiated ART.
Female self-report of adherence to antiretroviral treatment | Enrollment to 6 weeks, 14 weeks, and 6 months postpartum
  Women who report initiation of ART will be asked report on their degree of adherence to ART on a visual analogue scale.
Female self-report of infant mortality | Delivery to 6 weeks, 14 weeks, and 6 months postpartum
  At follow-up interviews, women will be asked to report whether the child they delivered was still alive.

OTHER OUTCOMES:
Incremental cost per pregnant woman enrolled | Enrollment to 6 months postpartum
Incremental cost-effectiveness per infant HIV infection averted | Enrollment to 6 months postpartum
Incremental cost-effectiveness per maternal HIV infection averted | Enrollment to 6 months postpartum
Incremental cost-effectiveness HIV-related death and disability adjusted life-year (DALY) averted | Enrollment to 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Carey Farquhar, MD MPH, Principal Investigator — University of Washington; Daisy Krakowiak, MPH, Study Director — University of Washington
Locations (1):
- Kisumu District Hospital, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Krakowiak D, Makabong'o P, Goyette M, Kinuthia J, Osoti AO, Asila V, Gone MA, Mark J, Farquhar C. Reaching hard-to-reach men through home-based couple HIV testing among pregnant women and their male partners in western Kenya: a qualitative study. BMC Public Health. 2020 May 19;20(1):724. doi: 10.1186/s12889-020-08878-0. PMID 32429879
- [Derived] Krakowiak D, Kinuthia J, Osoti AO, Asila V, Gone MA, Mark J, Betz B, Parikh S, Sharma M, Barnabas R, Farquhar C. Home-Based HIV Testing Among Pregnant Couples Increases Partner Testing and Identification of Serodiscordant Partnerships. J Acquir Immune Defic Syndr. 2016 Aug 1;72 Suppl 2(Suppl 2):S167-73. doi: 10.1097/QAI.0000000000001053. PMID 27355505